CLINICAL TRIAL: NCT02054715
Title: Evaluation of Psychoeducation for Cancer Patients Eligible for Clinical Trials
Brief Title: Multimedia Psychoeducation or Print Education in Preparing Cancer Patients for Decision Making About Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URCC12107; NCI-2013-02237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC12107 (Other: University of Rochester); URCC-12107 (Other: DCP); U10CA037420 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (print educational) (Experimental): Participants undergo a print educational intervention during which they meet with a site coordinator and are instructed to read the NCI booklet titled Taking Part in Cancer Treatment Studies, comprised primarily of information about the nature and conduct of cancer clinical trials.
  Interventions: Behavioral: print educational intervention
- Arm II (multimedia psychoeducational) (Experimental): Participants undergo a multimedia psychoeducational intervention during which they meet with a site coordinator and are instructed to view a DVD and read a booklet titled Clinical Trials: Are They Right For You? Participants are encouraged to watch the DVD and read the booklet again at home.
  Interventions: Behavioral: multimedia psychoeducational intervention

INTERVENTIONS:
Behavioral: print educational intervention — print educational intervention
  Other Names: intervention, educational
  Arms: Arm I (print educational)
Behavioral: multimedia psychoeducational intervention — multimedia psychoeducational intervention
  Other Names: intervention, educational
  Arms: Arm II (multimedia psychoeducational)

SUMMARY:
This randomized clinical trial compares multimedia psychoeducation to print education in preparing patients with cancer for decision making about clinical trial participation. Multimedia psychoeducation includes a digital video disc (DVD) and written materials with a combined focus on knowledge and attitude change, and may be an effective method to help patients prepare for decision making about clinical trial participation. It is not yet known whether a multimedia psychoeducation is more effective than print education in preparing patients for decision making about clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of intervention assignment on patients' preparedness for decision making about clinical trial participation.

SECONDARY OBJECTIVES:

I. To determine the effect of intervention assignment on indicators of the quality of patients' decision making about clinical trial participation.

II. To examine mechanisms by which multimedia psychoeducation (MP) exerts its expected positive effects on preparedness for decision making.

TERTIARY OBJECTIVES:

I. To explore the effects of intervention assignment on clinical trial participation.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants undergo a print educational intervention during which they meet with a site coordinator and are instructed to read the National Cancer Institute (NCI) booklet titled Taking Part in Cancer Treatment Studies, comprised primarily of information about the nature and conduct of cancer clinical trials.

ARM II: Participants undergo a multimedia psychoeducational intervention during which they meet with a site coordinator and are instructed to view a digital video disk (DVD) and read a booklet titled Clinical Trials: Are They Right For You? Participants are encouraged to watch the DVD and read the booklet again at home.

After completion of study, patients are followed up at 3-7 and 49-56 days.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak and read English
* Be diagnosed with cancer
* Have been informed of their eligibility for a specific phase II or III therapeutic clinical trial open for enrollment at the participating NCI Community Oncology Research Program (NCORP) site
* Have already met one or more eligibility criteria and have a reasonable expectation of meeting any remaining eligibility criteria for the therapeutic clinical trial
* Be capable of providing written informed consent for study participation

Exclusion Criteria:

* Participants must not have been asked previously to participate in another therapeutic cancer clinical trial
* Participants must not have already made a decision to participate in the phase II or III therapeutic clinical trial for which they were informed of their eligibility
* Participants must not have documented or observable visual, auditory, psychiatric, or neurological disorders that would interfere with study participation (e.g., blindness, deafness, psychosis, or dementia)
* Participants must not be eligible only for phase I trial; these patients are excluded because few of these trials are offered at NCORP sites and because their design and goals differ considerably from those of phase II and III trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Jacobsen, Principal Investigator — University of Rochester
Locations (18):
- United States (18):
  - San Diego State University, San Diego, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Hawaii MU-NCORP, Honolulu, Hawaii
  - Heartland NCORP, Decatur, Illinois
  - Kansas City Clinical Oncology Program, Prairie Village, Kansas
  - Gulf South MU-NCORP, New Orleans, Louisiana
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Metro MN NCORP, Minneapolis, Minnesota
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Nevada NCORP, Las Vegas, Nevada
  - URCC / University of Rochester NCORP Research Base, Rochester, New York
  - Southeast Clinical Oncology Research Consortium, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Dayton Community Oncology Program, Dayton, Ohio
  - Geisinger Cancer Institute NCORP, Danville, Pennsylvania
  - Greenville Health System Cancer Instutite/Greenville NCORP, Greenville, South Carolina
  - Wisconsin NCORP, Marshfield, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/publications/pdq

RESULTS

PARTICIPANT FLOW:
Period: Baseline/Follow-up 1
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Started | 219 | 199
Completed | 211 | 192
Not Completed | 8 | 7
Not completed — Refused | 1 | 3
Not completed — Medical | 0 | 1
Not completed — Changed MD/Facility | 0 | 1
Not completed — Disliked Procedure | 0 | 1
Not completed — No Reason | 0 | 1
Not completed — Overwhelmed | 2 | 0
Not completed — Ineligible | 3 | 0
Not completed — Hospitalization | 1 | 0
Not completed — Changed Mind | 1 | 0
Period: Follow-up 2
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Started | 211 | 192
Completed | 192 | 173
Not Completed | 19 | 19
Not completed — Lost to Followup | 3 | 1
Not completed — Refused | 3 | 2
Not completed — Followup Not Completed | 3 | 4
Not completed — Ineligible | 4 | 5
Not completed — Death | 3 | 3
Not completed — Hospitalization | 0 | 2
Not completed — Changed MD/Facility | 0 | 1
Not completed — Changed Mind | 0 | 1
Not completed — No Reason | 2 | 0
Not completed — Treatment Change or Delay | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational) | Total
Number analyzed (Participants) | 219 | 199 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.2) | 61.5 (12.6) | 61.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 121 | 255
  Male | 85 | 78 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 214 | 192 | 406
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 19 | 37
  White | 195 | 177 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Marital Status [Count of Participants; unit: Participants]
  Never Married | 19 | 20 | 39
  Currently Married | 133 | 113 | 246
  Separated | 9 | 4 | 13
  Divorced | 38 | 34 | 72
  Widowed | 18 | 28 | 46
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Preparedness for Decision Making About Clinical Trial Participation, Measured Using Scores From the Preparation for Decision Making Scale
Description: Preparation for Decision Making Scale (PDMS) is a valid and reliable 10-item self-report measure for which respondents rate the usefulness of materials they were provided in preparing them to communicate with their health care provider and make a health care decision. Each item is scored 1 to 5 where 1=Not at All, 2=A Little, 3=Somewhat, 4=Quite a Bit, 5=A Great Deal. Larger number is better. All 10 scores are summed, then divided by 10; The result - 1 is then multiplied by 25 and we have a range from 0 (less prepared) - 100 (most prepared).
Time Frame: Day 3 to 7
Population: There were 219 (PE) + 199 (MP) = 418 at Baseline. The population for this outcome is 211 (PE) + 192 (MP) = 403 This is defined as follow-up 1 (Day 3-7).
Measure: Mean (Standard Error); unit: percentage of PDMS (0 - 100)
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Number analyzed (Participants) | 211 | 192
percentage of PDMS (0 - 100) | 71.3 (1.4) | 71.2 (1.5)
Statistical Analysis 1: Comparison: Arm I (Print Educational) vs Arm II (Multimedia Psychoeducational); Two-sided F-Test as a statistical comparing MP and PE means; Test type: Other; p = 0.9621, F-Test; Mean Difference (MP - PE) = -0.10, 95% CI 2-sided [-4.1 to 3.9], Standard Error of Mean 2.0

2. Secondary Outcome: The Decision Regret Scale (DRS)
Description: The Decision Regret Scale (DRS) is a five-item paper and pencil self-report measure that asks subjects to reflect on a particular decision and then rate each item on a Likert scale from 1 (strongly agree) to 5 (strongly disagree). A mean score for the DRS is calculated by reverse scoring the two negatively phrased items and dividing by five. The mean scores are converted to a score ranging from 0 to 100 by subtracting 1 and multiplying by 25 and higher scores represent increases in the severity of decision regret. Higher scores are worse.
Time Frame: Day 49-56
Population: The population for this outcome is 192 (PE) + 173 (MP) = 365 This is defined as follow-up 2 (Day 49-56).
Measure: Mean (Standard Error); unit: percentage of DRS (0 - 100)
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Number analyzed (Participants) | 192 | 173
percentage of DRS (0 - 100) | 18.1 (1.1) | 18.3 (1.1)
Statistical Analysis 1: Comparison: Arm I (Print Educational) vs Arm II (Multimedia Psychoeducational); Two-sided F-Test comparing the MP and PE means; Test type: Other; p = 0.9065, F-test; Mean Difference (MP - PE) = 0.18, 95% CI 2-sided [-2.89 to 3.26], Standard Error of Mean 1.57

3. Secondary Outcome: The Decisional Conflict Scale (DCS)
Description: The Decisional Conflict Scale (DCS) is a valid and reliable 16-item self-report measure that assesses the extent to which respondents experience certainty, satisfaction, and confidence following a health care decision. In the present study, it will be keyed to the decision about therapeutic clinical trial participation. Instructions given to respondents include asking them to reflect on the decisions have just made or are about to make and to respond to statements in the DCS using a five-point Likert scale. Responses to each statement are scored from 1 (strongly agree) to 5 (strongly disagree), with negative statements having reverse scoring; thus high scores indicate higher decisional conflict.
Time Frame: Day 49-56
Population: The population for this outcome is 192 (PE) + 173 (MP) = 365 This is defined as follow-up 2 (Day 49-56).
Measure: Mean (Standard Error); unit: Percentage of DCS (0 - 100)
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Number analyzed (Participants) | 192 | 173
Percentage of DCS (0 - 100) | 18.0 (0.9) | 17.9 (1.1)
Statistical Analysis 1: Comparison: Arm I (Print Educational) vs Arm II (Multimedia Psychoeducational); Two-sided F-Test comparing the MP and PE means; Test type: Other; p = 0.9709, F-Test; Mean Difference (MP - PE) = -0.05, 95% CI 2-sided [-2.79 to 2.69], Standard Error of Mean 1.40

4. Other Pre Specified Outcome: To Explore the Effects of Intervention Assignment on Clinical Trial Participation.
Description: Given the ethical perspective that patients have a right to make autonomous decisions about clinical trial participation, no hypothesis is offered about the effect of intervention assignment on clinical trial participation rates. To conduct the exploratory analysis regarding the effects of intervention assignment on clinical trial participation, data for all patients offered participation in a therapeutic clinical trial will be entered into a 2 (Intervention: MP or PE) x 2 (Clinical Trial Participation: Yes or No/Still Deciding) contingency table and analyzed using either a Fisher exact test or chi-square test as appropriate.
Time Frame: Day 49-56
Population: The population for this outcome is 192 (PE) + 170 (MP) = 362 Note: There were 3 individuals (MP) who did not answer this question. This is defined as follow-up 2 (Day 49-56).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
Number analyzed (Participants) | 192 | 170
Participants
  Yes | 119 | 117
  No | 69 | 42
  Still Deciding | 4 | 11
Statistical Analysis 1: Comparison: Arm I (Print Educational) vs Arm II (Multimedia Psychoeducational); Chi-square test between MP and PE. 69% of subjects that got the Multimedia Psychoeducation intervention chose to participate in a clinical trial, compared with 62% in the Print Education group; Test type: Other; p = 0.014, Chi-squared

ADVERSE EVENTS:
Arm/Group | Arm I (Print Educational) | Arm II (Multimedia Psychoeducational)
All-Cause Mortality (participants affected / at risk) | 3/219 | 3/199
Serious Adverse Events (participants affected / at risk) | 4/219 | 3/199
Other Adverse Events (participants affected / at risk) | 1/219 | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Print Educational) (N=219) | Arm II (Multimedia Psychoeducational) (N=199)
Hyponatremia, decreased WBC, post chemo (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
metastatic hepatocellular carcinoma (Hepatobiliary disorders) | 1 (1) | 0 (0) — Death
Perirectal abscess, large tumor with post obstructive atelectasis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Death
Extensive metastatic melanoma (to skeletal system, liver, lungs, adrenal glands, mesentery, heart) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Death
Metastatic melanoma to liver/ sepsis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Death
Stage IV lung cancer with widespread mets (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Death
Death (General disorders) | 0 (0) | 1 (1) — Death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Print Educational) (N=219) | Arm II (Multimedia Psychoeducational) (N=199)
Fever post chemo (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

https://nctn-data-archive.nci.nih.gov/